CLINICAL TRIAL: NCT01430364
Title: BIfurcation Optimal Treatment Strategy With LIMus Eluting Dedicated Bifurcation Versus Convention Stent Randomized Study
Brief Title: BIfurcation Optimal Treatment Strategy With LYMus Eluting Dedicated Bifurcation Versus Convention Stent Randomized Study
Acronym: BIOSS LIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medica Cor Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSS LIM
Record Dates: First submitted 2011-09-03; First posted 2011-09-08 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Bifurcation Stenosis
Keywords: coronary bifurcation stenosis; dedicated bifurcation stent; sirolymus; PTS; BiOSS Lym

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIOSS implantation (Active Comparator)
  Interventions: Device: BIOSS LIM implantation; Device: BIOSS Lim; Device: CarloS

INTERVENTIONS:
Device: BIOSS LIM implantation — BIOSS LIM is a dedicated bifurcation stent system with sirolymus elution.
Device: BIOSS Lim
Device: CarloS

SUMMARY:
Study aims: to compare two intervention strategies for bifurcation treatment - provisional T-stenting (PTS) with drug-eluting stent (sirolimus eluting), with kissing balloon inflation at the end of procedure - the best treatment strategy at the moment, with stenting of bifurcation lesions with dedicated bifurcation drug-eluting stent BiOSS Lym.

DETAILED DESCRIPTION:
The coronary bifurcation lesions pose a therapeutic problem with high rates of periprocedural complications, higher rates of in-stent restenosis and stent thrombosis. These are lesions where stenting is not superior in comparison to balloon angioplasty in regard to side branch. It was demonstrated many times, in literature and in daily practice, that angiographically high grade ostial side branch stenosis is not flow limiting and do not cause ischemia, therefore do not require treatment. From the other side, our own data with magnetic resonance imaging (MRI) before and after bifurcation percutaneous coronary intervention (PCI) demonstrated that occurrence of angiographic stenosis more than 70% in diameter is associated with periprocedural myonecrosis in the region of side branch. This fact puts a very important question about the mechanisms of this myonecrosis. If the jailed side branch has no significant flow limiting stenosis, but there is some degree of residual ischemia, which after some period of persistence could lead to myonecrosis, will mean that more aggressive treatment of ostial stenosis is needed. It is interesting that the strategy of treatment is very important, because techniques with second stent implantation (with primary purpose to limit side branch (SB) ischemia) are associated with higher grade of troponin increase. Of course this is association and not causality, despite that in randomized study it was confirmed also.

Even after the introduction of drug-eluting stents (DES) in the treatment of coronary bifurcation lesions, important basic problems remain. It was proposed that these problems are related to non-dedicated design of conventional stent intended for treatment of straight vessel segments. Thus any deformation of the stents during bifurcation implantation depends on the stent cell shape, size and material properties (11). To resolve these problems it was suggested to make dedicated bifurcation stents (1, 2, 11). However, the special "dedication" per se is not defined and unclear as terminology - the stent could be dedicated for patient fitting the anatomical characteristics of particular bifurcation point (vessel diameters, angulations), giving better hemodynamic conditions; or stent could be dedicated for operator to make the procedure quicker and safer, eliminating or limiting SB compromise. Probably the best option is the combination of both characteristics.

The currently available stents on the market generally target the second requirement. Three groups of stents are available at this moment - proximal main vessel (MV) stent (Axxess, Devax, USA), MV stenting across the SB with different designs making possible permanent access to SB and finally purely SB dedicated stents (Tryton, Sideguard, Biguard). Neither of these stents did not match proximal - distal MV size difference nor take into account between vessel angulations. The device success rate varies considerably (75% - 100%); however the study with 100% success was performed in only 11 patients. For all other devices the success rate is around 85%. The proximal MV stent and SB only stents require additional stent implantation for non-intended vessel. Stents designed to have permanent access to SB are implanted over 2 wires, which in reality makes the procedure more difficult and demanding rather to simplify it (which was the primary intention of those stents). The reasons are wires crisscrossing, wire-bias in proper orientation of device to SB (rotational and axial positioning). This, along with requirement of larger guide catheter size explains why the dedicated stents do not gain popularity in the interventional cardiology community.

The BiOSS Lim stent (Balton, Warsaw, Poland) is completely different from the above systems. The stent is designed to be user friendly: it tracked over one wire and its profile is quite low (1.08mm), which make it possible to implant it even through 5 Fr guiding catheter. The stent fits the bifurcation anatomy - it matches the proximal - distal diameters of the main vessel (MV); as it permits deformation in its mid-part it can adapt exactly on main vessel - main branch angle angle, making wide opening to SB. If the SB must be dilated the stent recrossing is very easy, because wider proximal and narrow distal parts give step-down at carina tip region, in this way self direct wire to SB. The proximal and distal parts of the stent work independently and SB could be safely dilated without need from kissing balloon inflation as no deformation of contralateral wall strut. This simplifies and shortens the procedure. And finally, the stent construction prevents carina displacement, as a basic mechanism of side branch compromise.

Study aims: to compare two intervention strategies for bifurcation treatment - provisional T-stenting (PTS) with drug-eluting stent (sirolimus eluting), with kissing balloon inflation at the end of procedure - the best treatment strategy at the moment, with stenting of bifurcation lesions with dedicated bifurcation drug-eluting stent BiOSS Lym.

ELIGIBILITY:
1. Inclusion Criteria

   * Subject at least 18 years of age.
   * Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
   * Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
   * Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.
2. Exclusion Criteria

   * STEMI
   * Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
   * Subjects who refuse to give informed consent.
   * Subjects with LVEF<30%
   * Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy
   * Contraindications for 12 months DAP

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 12 months
  death, myocardial infarction (MI), target vessel revascularization (TVR)

SECONDARY OUTCOMES:
Target lesion revascularization (TLR) | 12 months
  Clinically driven revascularization rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Medica Cor Heart Hospital, Rousse, Bulgaria